CLINICAL TRIAL: NCT00248976
Title: Improving Health Behavior and Outcomes After Angioplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Mary E. Charlson, MD, The William T. Foley Distinguished Professor in Medicine, Weill Medical College of Cornell University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0698-267
Record Dates: First submitted 2005-11-03; First posted 2005-11-04 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Angioplasty
Keywords: Angioplasty; Motivating behavior change; Reducing risk factors; Enhancing quality of life; Improving treatment outcomes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): This is the control group, which will be monitor. No intervention will be delivered to this group.
- 2 (Experimental): This group received the experimental intervention. This is an intervention based on feedback of individualized risk profiles framed as the opportunity to reduce one's biologic age. Net-present value of individual health behaviors in years.
  Interventions: Behavioral: Net-present value of individual health behaviors in years

INTERVENTIONS:
Behavioral: Net-present value of individual health behaviors in years
  Arms: 2

SUMMARY:
The objective of this randomized trials is to evaluate, among coronary artery disease patients who have just had either angioplasty or stents, whether a novel intervention based on feedback of individualized risk profiles framed as the opportunity to reduce one's biological age is more effective after two years in reducing mortality and major cardiovascular morbidity (specifically, myocardial infarction, stroke, class II-IV angina, and severe ischemia) than the standard risk reduction approach, which is framed as one's opportunity to reduce future risk. The novel strategy is based on the theory of net-present value and is tested in coronary artery disease patients who have a high risk of adverse outcomes by two years.

DETAILED DESCRIPTION:
1. To determine whether patients who receive the net-present value intervention have more improvements in their risk factor profile than those in the control group at two years.
2. To determine whether the net-present value intervention will enable patients to sustain behavioral change over the long-term.
3. To determine whether the net-present value intervention will improve overall functional status and prevent further disability.

The long-term objective of this study is to determine whether a net-present value approach for motivation behavior change is effective in reducing risk factors, improving treatment outcomes, and enhancing quality of life among a high-risk group of patients.

ELIGIBILITY:
Inclusion criteria:

* All patients undergoing coronary artery catheterization who are found to have at least single vessel stenosis and who have had revascularization with angioplasty or coronary artery stenting will be eligible for enrollment. Patients must be able to provide informed consent within the one week after the procedures.

Exclusion criteria:

* Patients must be verbally fluent in English. To ascertain this, we ask the patient to rate their fluency on a scale of 1-10 (with 10 as best), and if the score is 7 or more, they are approached for consent. The patient must be able to provide their own consent without translation.
* Enrollment in other trials designed to modify post-procedure behaviors.
* Patients who refuse to participate will be excluded.
* If at any time prior to enrollment in the study, the patient's cardiologist determines that the patient should not participate in this study, the patient will not be enrolled in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 1999-04; Primary Completion 2004-03-29 (Actual); Study Completion 2004-03-29 (Actual)

PRIMARY OUTCOMES:
Mortality
Myocardial Infarction
Angina
Severe ischemia on non-invasive testing
Stroke

SECONDARY OUTCOMES:
a. To determine whether patients who receive the net-present value intervention have more improvements in their risk factor profile than those in the control group at two years.
b. To determine whether the net-present value intervention will enable patients to sustain behavioral change over the long-term.
c. To determine whether the net-present value intervention will improve overall functional status and prevent further disability.

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Charlson, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- New York Presbyterian College-Weill Medical Center, New York, New York, United States